CLINICAL TRIAL: NCT00319449
Title: A Single Center, Randomized, Parallel Groups, Placebo-Controlled Study Comparing The Efficacy, Safety, And Tolerability Of The Daily Co-administration Of Ezetimibe 10 Mg Or Ezetimibe Placebo To Ongoing Treatment With Atorvastatin 10 Mg In Subjects With Primary Hypercholesterolemia And Multiple Coronary Heart Disease Risk Factors in Indonesian Population.
Brief Title: Adding Ezetimibe Tablet to Ongoing Treatment With Atorvastatin in Subjects With High Cholesterol and Multiple Coronary Heart Disease Risk Factors (Study P04060)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: PT. Schering-Plough. Tbk Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04060
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Coronary Arteriosclerosis
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Ezetimibe 10 mg (Experimental): Participants treated with 10 mg/day ezetimibe added to an ongoing treatment of 10 mg/day atorvastatin.
  Interventions: Drug: Ezetimibe; Drug: Atorvastatin 10 mg
- Placebo 10 mg (Placebo Comparator): Participants treated with 10 mg/day matching placebo to ezetimibe added to an ongoing treatment of 10 mg/day atorvastatin.
  Interventions: Drug: Placebo; Drug: Atorvastatin 10 mg

INTERVENTIONS:
Drug: Ezetimibe — 10 mg ezetimibe, orally, daily for 6 weeks, added to ongoing treatment with 10 mg atorvastatin
  Arms: Ezetimibe 10 mg
Drug: Placebo — 10 mg/day matching placebo to ezetimibe, orally, daily for 6 weeks, added to ongoing 10 mg atorvastatin
  Arms: Placebo 10 mg
Drug: Atorvastatin 10 mg — 10 mg/day atorvastatin, orally, (ongoing treatment in participants)

SUMMARY:
This study is being conducted to compare the efficacy, safety, and tolerability of ezetimibe 10 mg coadministered with atorvastatin 10 mg versus atorvastatin 10 mg in Indonesian population with primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an LDL-C concentration >= 3.3 mmol/L (130 mg/dL) to <= 4.9 mmol/L (190 mg/dL) using the Freidewald calculation.
* Participants must have triglyceride concentrations of < 3.99 mmol/L (350 mg/dL).
* Participants must have two or more coronary heart disease risk factors listed below:

  * Current cigarette smoking
  * Hypertension (BP >= 140/90 mmHg or on antihypertensive medication)
  * Low HDL cholesterol (< 40 mg/dL)
  * Family history of premature CHD (CHD in male first degree relative < 55 years; CHD in female first degree relative < 65 years)
  * Age (Men >= 45 years; women >= 55 years)
* Participant must be currently taking atorvastatin 10 mg daily and by history has taken 80% of daily doses for the 6 weeks prior to participating.
* Participants must have liver transaminases (ALT, AST) < 50% above the upper limit of normal, with no active liver disease, and CK < 50% above the upper limit of normal.
* Participants must have maintained a cholesterol lowering diet, exercise program, and stable weight for at least 4 weeks prior to the study and be willing to continue the same diet and exercise program during the study.
* Women receiving hormonal therapy, including hormone replacement, any estrogen antagonist/agonist, or oral contraceptives, must have been maintained on a stable dose and regimen for at least 8 weeks and be willing to continue the same regimen for the duration of the study.

Exclusion Criteria:

* Participants who meet any of the following criteria will be excluded:
* Body mass index (BMI = weight [kg]/height**2[m]) is >= 30 Kg/m**2.
* Consume > 14 alcoholic drinks per week.
* Women who are pregnant or nursing.
* Congestive heart failure defined by NYHA as Class III or IV.
* Uncontrolled cardiac arrhythmia.
* Coronary heart disease (CHD).
* Unstable or severe peripheral artery disease within 3 months of participating
* Uncontrolled hypertension (treated or untreated) with systolic blood pressure > 160 mm Hg or diastolic > 100 mm Hg.
* Type I or Type II diabetes mellitus.
* Secondary causes of hyperlipidemia, such as secondary hypercholesterolemia due to hypothyroidism.
* Impaired renal function (creatinine > 2.0 mg/dL) or nephrotic syndrome.
* Known HIV positive.
* Cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas).
* History of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.
* Participants who are on any of the following concomitant medications:
* Participants who are on medications that are potent inhibitors of CYP3A4, including cyclosporine, systemic itraconazole, fluconazole, and ketoconazole, erythromycin or clarithromycin, nefazodone, mibefradil, protease inhibitors and large amounts of grapefruit juice (> 1 quart/day).
* Participants who are on lipid-lowering agents (other atorvastatin): niacin (> 200 mg/day)
* Participants who are on over the counter lipid lowering agents such as fish oils, garlic and cholestin
* Participants who are on oral corticosteroids, unless used as replacement therapy for pituitary/adrenal disease and the subject is on a stable regimen for at least 6 weeks.
* Participants who are currently using psyllium, other fiber-based laxatives, and/or any other OTC therapy known to affect serum lipid levels (phytosterol margarine), and have not been on a stable regimen for at least 5 weeks and who do not agree to remain on this regimen throughout the study.
* Participant who are currently using orlistat or sibutramine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ezetimibe 10 mg | Placebo 10 mg
Started | 10 | 12
Completed | 8 | 12
Not Completed | 2 | 0
Not completed — Subject did not wish to continue | 1 | 0
Not completed — Noncompliance with the protocol | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe 10 mg | Placebo 10 mg | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (12.1) | 52.2 (10.4) | 54.5 (11.3)
Age, Customized [Number; unit: Participants]
  18 to <65 years | 7 | 11 | 18
  65 or older | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  Indonesia | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Low Density Lipoprotein-cholesterol (LDL-C) at Baseline and After 6 Weeks of Treatment With Ezetimibe 10 mg Added to Atorvastatin 10 mg Versus Placebo Added to Atorvastatin 10 mg
Description: 12-hour fasting blood samples were collected in participants to measure high density lipoprotein-cholesterol (HDL-C), triglycerides and total cholesterol. LDL-C was measured using Friedewald calculation (LDL-C = Total C - [HDL-C + TG/5]) before and after treatment.
Time Frame: Baseline and 6 weeks
Population: Participants who completed the study.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ezetimibe 10 mg | Placebo 10 mg
Number analyzed (Participants) | 8 | 12
mg/dL
  Baseline | 148.125 [130.126 to 166.124] | 151.083 [136.387 to 165.780]
  6 weeks post treatment | 106.000 [89.030 to 122.970] | 108.273 [92.923 to 123.622]

2. Secondary Outcome: Number of Participants Who Achieve the Target LDL-C Concentration of < 3.3 mmol/L (130 mg/dL)
Description: 12-hour fasting blood samples were collected in participants to measure high density lipoprotein-cholesterol (HDL-C), triglycerides and total cholesterol. LDL-C was measured using Friedewald calculation (LDL-C = Total C - [HDL-C + TG/5] after treatment for 6 weeks.
Time Frame: 6 weeks post treatment
Population: Participants who completed the study.
Measure: Number; unit: Participants
Arm/Group | Ezetimibe 10 mg | Placebo 10 mg
Number analyzed (Participants) | 8 | 12
Participants | 7 | 8

3. Secondary Outcome: High Density Lipoprotein-cholesterol (HDL-C), Total Cholesterol and Triglycerides at Baseline and After 6 Weeks of Treatment With Ezetimibe 10 mg Added to Atorvastatin 10 mg Versus Placebo Added to Atorvastatin 10 mg
Description: 12-hour fasting blood samples were collected in participants and the high density lipoprotein-cholesterol (HDL-C), triglycerides and total cholesterol was measured with the basic lipid panel test.
Time Frame: 6 weeks post treatment
Population: Participants who completed the study.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ezetimibe 10 mg | Placebo 10 mg
Number analyzed (Participants) | 8 | 12
mg/dL
  HDL-C at baseline | 53.250 [44.579 to 61.921] | 57.667 [50.586 to 67.747]
  HDL-C at 6 weeks | 52.625 [43.954 to 61.296] | 53.500 [46.420 to 60.580]
  Total Cholesterol at baseline | 219.125 [202.355 to 235.895] | 226.000 [212.307 to 239.693]
  Total Cholesterol at 6 weeks | 156.375 [139.605 to 173.145] | 185.667 [171.974 to 199.359]
  Triglycerides at baseline | 139.500 [105.213 to 173.787] | 131.667 [103.672 to 159.662]
  Triglycerides at 6 weeks | 115.250 [80.963 to 149.537] | 120.250 [92.255 to 148.245]

ADVERSE EVENTS:
Arm/Group | Ezetimibe 10 mg | Placebo 10 mg
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/12
Other Adverse Events (participants affected / at risk) | 2/10 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ezetimibe 10 mg (N=10) | Placebo 10 mg (N=12)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ezetimibe 10 mg (N=10) | Placebo 10 mg (N=12)
Nausea (Gastrointestinal disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
pruritis (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Protocol deviations may have occurred that resulted in quality issues associated with reporting of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator (PI) agrees not to publish or publicly present

any interim results of the Study without prior written consent of the SPONSOR.

The PI further agrees to provide thirty (30) days written notice to the SPONSOR prior to submission for publication or presentation to allow SPONSOR to review abstracts or manuscripts for publication.